CLINICAL TRIAL: NCT00595257
Title: Feasibility Study of the Safety and Activity of Autologous Bone Marrow Aspirate Concentrate (BMAC) for the Treatment of Non Reconstructable Critical Limb Ischemia Due to Peripheral Arterial Occlusive Disease
Brief Title: Feasability Study of Autologous Bone Marrow Aspirate Concentrate for Treatment of CLI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Harvest Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TriCell/CT/IND-001
Record Dates: First submitted 2007-12-19; First posted 2008-01-16 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Arterial Occlusive Diseases
Keywords: PAD, CLI, Critical Limb Ischemia, bone marrow, stem cell, injection, infusion
MeSH Terms: conditions — Arterial Occlusive Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): injection of BMAC into ischemic limb
  Interventions: Device: centrifuge, laboratory, tabletop (SmartPReP2 BMAC System)
- 2 (Active Comparator): Injection and Infusion of BMAC into ischemic lower limb
  Interventions: Device: centrifuge, laboratory, tabletop (SmartPReP2 BMAC System)

INTERVENTIONS:
Device: centrifuge, laboratory, tabletop (SmartPReP2 BMAC System) — autologous bone marrow aspirate will be concentrated using the SmartPRep2 BMAC system and then injected/infused into ischemic limbs
  Other Names: SmartPReP2 BMAC System

SUMMARY:
The purpose of this study is to determine if concentrated nucleated cells from your own bone marrow, injected or infused into an ischemic limb, will restore sufficient blood flow to avoid amputation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Critical Limb Ischemia per protocol (see diagnostic criteria #2) with regard to the study limb.

   Existence of a PAOD with clinical presentation corresponding to Rutherford Category 4 or Category 5 as defined in the reporting standards adopted by the Society of Vascular Surgeons (table 1)
2. Patient meets at least one of the following diagnostic criteria in the study limb:

   * Ankle artery occlusion pressure absolute <50 mmHg or ABI <0.4
   * Toe artery occlusive pressure < 40mm Hg or TBI (<0.4)
   * TcPO2 <20 mmHg lying down breathing room air, if available.
3. There is no reasonable open surgical or endovascular revascularization option as determined by the treating vascular specialist. Factors that may contribute to the determination of inoperability may include:

   * Anatomical considerations

     * No outflow targets
     * No appropriate conduit (i.e. vein for bypass)
     * Long segment occlusions or calcified lesions that predict poor outcome with endovascular approaches.
   * High risk medical conditions

     * Unstable cardiac disease.
     * Renal insufficiency
   * History of prior failed revascularization attempts
   * The patient's unsuitability must be confirmed by 2 qualified physicians.

     * The attending vascular surgeon will provide the primary assessment.
     * The confirmatory opinion must come from a fully licensed physician. (not a resident)
     * If anatomical considerations are invoked, the second physician may be a vascular surgeon, interventional radiologist, cardiologist, or vascular medicine specialist.
     * If medical co-morbidity is deemed the high risk aspect, then the confirmatory opinion may be obtained from an internist, family physician, cardiologist, vascular medicine, nephrologists, or vascular surgeon.
4. Age >18 years and ability to understand the planned treatment
5. Subject has read and signed the IRB/IEC approved Informed Consent form
6. Patients for whom the following medication(s) is prescribed must have a one month stable baseline of appropriate/maximally tolerated therapy prior to enrollment: Plavix/asprin therapy, anticoagulation therapy, cholesterol lowering agent, and or blood pressure medication
7. Hematocrit ≥ 28.0%, White Blood Cell count ≤ 14,000, Platelet count ≥ 50,000, INR ≤ 1.6 unless on Coumadin, or PTT <1.5 x control (to avoid bleeding complications) Patients on Coumadin will be corrected prior to the procedure and must have an INR<1.6 at the time of randomization/surgery.

Exclusion Criteria:

1. Life expectancy <6 months due to concomitant illnesses
2. History of bone marrow diseases (especially NHL, MDS) that prohibit transplantation
3. Terminal renal failure with existing dependence on dialysis
4. Known active malignancy or results outside of normal limits from the following tests: PAP, Chest X-ray, PSA, Mammogram, Hemocult unless follow-up studies reveal patient to be cancer free..
5. Poorly controlled diabetes mellitus (HgbA1C>10%)
6. Medical risk that precludes anesthesia (conscious sedation), or ASA Class 5
7. Life-threatening complications of the ischemia necessitating immediate amputation
8. Uncorrected iliac artery occlusion on index side
9. Extensive necrosis of the index limb or other conditions that make amputation inevitable (Rutherford Category 6)
10. Active clinical infection being treated by antibiotics within one week of enrollment
11. Treatment with immunosuppressant drugs (including Prednisone > 5 mg per day).
12. Female who is pregnant or nursing, or of child bearing potential and is not using a reliable birth control method.
13. Underwent a major cardiovascular surgical procedure (carotid endarterectomy, open arterial aneurysm or bypass surgery, or coronary artery bypass surgery) or an adverse cardiovascular event (stroke or MI) within the 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
avoid amputation | 60 days

SECONDARY OUTCOMES:
measurement of hemodynamic response | 60 Days

CONTACTS AND LOCATIONS:
Overall Officials: R E Arasan, MD, Study Director — LifeCell India
Locations (1):
- Sri Ramachandra University Medical Center, Porur, Chennai, India